CLINICAL TRIAL: NCT00038688
Title: A Phase III Randomized Study to Evaluate the Efficacy of a Network-Oriented Peer Education Intervention for the Prevention of HIV Transmission Among Injection Drug Users and Their Network Members
Brief Title: A Study of Peer Education to Prevent HIV Transmission Among Injection Drug Users and Their HIV Risk Contacts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 037
Record Dates: First submitted 2002-06-04; First posted 2002-06-05 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2006-03

CONDITIONS: HIV Infections
Keywords: Health Education; Substance Abuse, Intravenous; Program Evaluation; Peer Group; Risk-Taking; HIV Seronegativity; Substance-related Disorders
MeSH Terms: conditions — HIV Infections; Health Education; Substance Abuse, Intravenous; Risk-Taking; Substance-Related Disorders

INTERVENTIONS:
Behavioral: Peer HIV Education Program

SUMMARY:
Injection drug use is the major mode of HIV transmission in many countries. Injection drug users (IDUs) transmit HIV not only through shared drug injection equipment but also through heterosexual and homosexual transmission and mother-to-child transmission. Studies have shown that peer education programs can reduce HIV risk behavior in IDUs. However, it is not known if reduced HIV risk behavior leads to fewer HIV infections. The purpose of this study is to find out if a peer education program can reduce the number of new HIV infections by changing the behavior of IDUs and their HIV risk contacts.

DETAILED DESCRIPTION:
More than 20 years of research in implementing interventions for IDUs indicate that HIV transmission among these users can be prevented, slowed, and stopped with the appropriate intervention. Intervening early with multiple strategies can prevent epidemic spread and its consequences. Even after prevalence has increased substantially, prevention interventions can reduce the further spread of HIV in drug-using populations and transmission into other populations. Although research results have been promising, it is unknown if self-reported behavior change is correlated with reducing rates of HIV transmission. This study will determine the efficacy of a peer-educator, network-oriented intervention to prevent HIV transmission among substance users and their risk network members. IDUs will be recruited using street and community outreach methods in Chiang Mai and Chiang Rai, Thailand and in Philadelphia, Pennsylvania, USA.

Individuals at the study clinics will undergo a screening survey and HIV counseling and testing; they will return to the clinic to receive their HIV test results, post-test counseling, and further screening. Those who are HIV uninfected, meet preliminary eligibility requirements, and are willing to participate will be enrolled as index participants. Each index participant will be asked to identify and attempt to recruit at least two other people (potential network members) whom he/she has had sex with or taken drugs with in the 3 months prior to screening. Infected and uninfected network members will be eligible for enrollment. Index participants will be randomly assigned with their network members to either the intervention group or a control group. All participants will receive HIV counseling and regular HIV testing. Index participants assigned to the intervention group attend six, two-hour peer educator-training sessions over a period of 4 weeks. The training sessions focus on skills building and promotion of risk-reducing behaviors. A one-hour booster training session is held for index participants after their 6- and 12-month follow-up assessments.

The study will last approximately 48 months, with enrollment expected to take about 30 months. Participants will be followed for a minimum of 18 months and a maximum of 30 months. Both index participants and network members have follow-up visits every 6 months, at which they will complete surveys designed to assess HIV risk behavior, network characteristics, the intensity of the intervention delivery, and social harms that may be associated with study participation. Average network HIV incidence rates will be compared for the two study groups.

NOTE: as of January 31, 2006, the HPTN 037 trial was terminated. Participants enrolled in the study will continue to be followed at a reduced number of study visits.

ELIGIBILITY:
NOTE: as of January 31, 2006, the HPTN 037 trial was terminated. Participants enrolled in the study will continue to be followed at a reduced number of study visits.

Inclusion Criteria for Index Participants

* HIV uninfected within 60 days of study entry
* Injected drugs at least 12 times in the last 3 months
* Out of methadone maintenance treatment for at least 3 months and have relapsed
* Willing to identify and attempt to recruit at least two HIV risk network members who are eligible for study
* Able to recruit at least one HIV risk network member eligible for study participation

Inclusion Criteria for Network Members

* Recruited by an eligible index participant for the study
* Have injected drugs with and/or had sex with the relevant index participant within 3 months prior to screening

Exclusion Criteria

* For index participants: prior or concurrent enrollment in another HIV behavioral or biomedical prevention study (e.g., vaccine or microbicide research, or any other behavioral or clinical research to test an intervention aimed at preventing or reducing the risk of HIV infection)
* Already enrolled in another network of HPTN 037 as a network member or index participant
* Mental, learning, or any other problems that would interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2610

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, PhD, Study Chair — Johns Hopkins Bloomberg School of Public Health, Johns Hopkins University
Locations (3):
- United States (2):
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - RAP Office, Philadelphia, Pennsylvania
- Research Institute for Health Sciences, Chiang Mai, Thailand

REFERENCES:
- [Background] Needle RH, Coyle SL, Normand J, Lambert E, Cesari H. HIV prevention with drug-using populations--current status and future prospects: introduction and overview. Public Health Rep. 1998 Jun;113 Suppl 1(Suppl 1):4-18. No abstract available. PMID 9722806
- [Background] Rietmeijer CA, Kane MS, Simons PZ, Corby NH, Wolitski RJ, Higgins DL, Judson FN, Cohn DL. Increasing the use of bleach and condoms among injecting drug users in Denver: outcomes of a targeted, community-level HIV prevention program. AIDS. 1996 Mar;10(3):291-8. PMID 8882669
- [Background] Latkin CA, Mandell W, Vlahov D, Oziemkowska M, Celentano DD. The long-term outcome of a personal network-oriented HIV prevention intervention for injection drug users: the SAFE Study. Am J Community Psychol. 1996 Jun;24(3):341-64. doi: 10.1007/BF02512026. PMID 8864208
- [Background] Kamb ML, Fishbein M, Douglas JM Jr, Rhodes F, Rogers J, Bolan G, Zenilman J, Hoxworth T, Malotte CK, Iatesta M, Kent C, Lentz A, Graziano S, Byers RH, Peterman TA. Efficacy of risk-reduction counseling to prevent human immunodeficiency virus and sexually transmitted diseases: a randomized controlled trial. Project RESPECT Study Group. JAMA. 1998 Oct 7;280(13):1161-7. doi: 10.1001/jama.280.13.1161. PMID 9777816
- [Background] Latkin CA, Sherman S, Knowlton A. HIV prevention among drug users: outcome of a network-oriented peer outreach intervention. Health Psychol. 2003 Jul;22(4):332-9. doi: 10.1037/0278-6133.22.4.332. PMID 12940388
- [Background] Latkin CA, Forman V, Knowlton A, Sherman S. Norms, social networks, and HIV-related risk behaviors among urban disadvantaged drug users. Soc Sci Med. 2003 Feb;56(3):465-76. doi: 10.1016/s0277-9536(02)00047-3. PMID 12570967
- [Derived] Hernandez-Ramirez RU, Spiegelman D, Lok JJ, Forastiere L, Friedman SR, Latkin CA, Vermund SH, Buchanan AL. Overall, Direct, Spillover, and Composite Effects of Components of a Peer-Driven Intervention Package on Injection Risk Behavior Among People Who Inject Drugs in the HPTN 037 Study. AIDS Behav. 2024 Jan;28(1):225-237. doi: 10.1007/s10461-023-04213-x. Epub 2023 Nov 7. PMID 37932493
- [Derived] Latkin C, Donnell D, Liu TY, Davey-Rothwell M, Celentano D, Metzger D. The dynamic relationship between social norms and behaviors: the results of an HIV prevention network intervention for injection drug users. Addiction. 2013 May;108(5):934-43. doi: 10.1111/add.12095. Epub 2013 Jan 30. PMID 23362861